CLINICAL TRIAL: NCT06235034
Title: Diagnostic CT Palliative Radiotherapy: Feasibility Study of Treating Bone Metastases
Brief Title: Diagnostic CT Palliative Radiotherapy: Feasibility Study of Treating Bone Metastases Without a CT Simulation
Acronym: dCT-PRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: dCT-PRT
Record Dates: First submitted 2023-12-21; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-12

CONDITIONS: Bone Metastases
Keywords: Palliative Radiation; CT Simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diagnostic CT (Experimental): patients will have their palliative radiotherapy designed on their diagnostic CT
  Interventions: Other: Diagnostic CT

INTERVENTIONS:
Other: Diagnostic CT — radiotherapy will be designed on diagnostic CT. If plan is of sufficient quality, RT will be delivered to patient

SUMMARY:
The purpose of this non-randomized, prospective study is to assess the feasibility of planning and delivering conventional palliative radiotherapy to bone metastases on previously available diagnostic CT scans (dCT).

Objectives:1) dosimetric accuracy of palliative radiotherapy designed on a dCT compared to a CT simulation 2) assess suitability of patient set up using surface landmarks and kilo voltage (kV) imaging 3) determine the proportion of patients who can receive radiotherapy designed on a dCT 4) confirm eligibility criteria for appropriate patients in clinical practice

All enrolled patients will undergo a CT simulation with tattoos as per current standard of care.The radiation oncologist will place fields on the dCT and CT simulation. Radiotherapy will be planned on both CT scans and reviewed for quality by both the radiation oncologist and medical physicist.

DETAILED DESCRIPTION:
Purpose:

This prospective study aims to demonstrate the feasibility of delivering palliative radiotherapy designed on a diagnostic CT scan (dCT) for patients with bone metastases in the spine and bony pelvis.

Hypothesis:

At least eighty percent of patients will successfully receive radiotherapy as designed on the dCT.

Justification:

Currently, patients who require palliative radiotherapy for bone metastases undergo a CT simulation and tattoos to design their radiotherapy. However, many of these patients already have a diagnostic CT scan. Other cancer centres have developed protocols to design radiotherapy on diagnostic CT scans. This technique allows patients to avoid CT simulations which can delay access treatment and can be burdensome for frail patients. The successful implementation of a diagnostic CT palliative radiotherapy (dCT-RT) workflow could provide more timely access to radiotherapy for patients, decrease resource utilization (CT simulation time, radiation therapist and nursing time), and decrease the carbon footprint of this service by decreasing the number of trips required to the cancer centre.

Objectives:

Primary: 1) dosimetric accuracy of palliative radiotherapy designed on a dCT compared to a CT simulation 2) assess suitability of patient set up using surface landmarks and kilo voltage (kV) imaging 3) determine the proportion of patients who can receive radiotherapy designed on a dCT 4) confirm eligibility criteria for appropriate patients in clinical practice

Secondary: 1) patient satisfaction with treatment process 2) evaluate carbon footprint savings of dCT-RT workflow

Research Design and Statistical Analysis:

This non-randomized prospective feasibility study will enroll ten eligible patients. All study activities will take place at BC Cancer, Vancouver Centre. Eligible patients will have their dCT reviewed by a radiation oncologist and medical physicist to determine suitability for radiotherapy planning. All enrolled patients will undergo a CT simulation with tattoos as per current standard of care. Radiotherapy will be planned on both their dCT scan and CT simulation. Patient set up will be performed using surface landmarks and confirmed with KV imaging. Quality assurance (QA) per the centres standard of practice will occur for plan review, approval and treatment set up. If at any point during the QA process accepted standards are not met, radiotherapy with be delivered according to the standard practice CT simulation plan.

Patient, tumor and treatment factors will be collected from the electronic medical record (Cerner) and radiotherapy plan in Aria and evaluated using descriptive statistics. Dosimetric parameters between dCT and CT simulation plans will be compared. The suitability of the dCT-RT plan will be documented as yes/no. The time required to set up a patient up for the dCT-RT workflow on day one will be record. Suitability of patient set up and deliverability of dCT-RTplan will be documented as yes/no. Patient satisfaction will be assessed post treatment with a brief questionnaire and described using descriptive statistics. The carbon footprint saved by the dCT-RT method will be calculated by assessing the carbon footprint associated with travel from home (or hospital) to the cancer centre.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Able to provide informed consent
* Patient able to lie supine comfortably
* Patient is receiving conventional palliative radiotherapy (Parallel Opposed Pair or single field over 8/1 or 20/5) for the treatment of bone metastases in the following locations: T5-lumbosacral spine, Bony pelvis
* Patient has a diagnostic CT scan which includes the anatomic location to be treated that is within 28 days of enrollment
* Quality of dCT scan is deemed sufficient for RT planning as determined by medical physicist and RT

Exclusion Criteria:

* Patient unwilling, unable to consent to treatment/study
* Any contraindications to receiving radiotherapy including pregnancy
* Oncologic emergencies, on call treatments, or any indications for urgent radiotherapy
* Inability to comfortably maintain and immobilized position due to uncontrolled pain or co-morbidities
* Cases requiring VMAT planning or complex planning to account for prior courses of radiotherapy
* Cases using non-conventional palliative radiotherapy fractionations
* Anatomic sites outside of the pre-defined criteria above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
dosimetric accuracy of palliative radiotherapy designed on a dCT compared to a CT simulation | 1 Year
assess suitability of patient set up using surface landmarks and kilo voltage (kV) imaging | 1 Year
determine the proportion of patients who can receive radiotherapy designed on a dCT | 1 Year
confirm eligibility criteria for appropriate patients in clinical practice | 1 Year

SECONDARY OUTCOMES:
patient satisfaction with treatment process | 1 Year
evaluate carbon footprint savings of dCT-RT workflow | 1 Year